CLINICAL TRIAL: NCT05924438
Title: Opti-DOR: A Randomised, Phase 3 Non-inferiority Study of DOR/3TC/TDF Compared to DTG/TAF/FTC in Participants Infected With HIV-1 Starting First-line Antiretroviral Therapy
Brief Title: A Randomised, Phase 3 Non-inferiority Study of DOR/3TC/TDF Compared to DTG/TAF/FTC in Participants Infected With HIV-1 Starting First-line Antiretroviral Therapy
Acronym: Opti-DOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Francois Venter (Other)
Collaborators: Africa Health Research Institute (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Professor Francois Venter, Professor, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZ-JW-033; DOH-27-052023-5232 (Other: South African National Clinical Trials Registry)
Record Dates: First submitted 2023-05-23; First posted 2023-06-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: HIV-1-infection
Keywords: delstrigo; KOCITAF; doravirine; HIV-1 RNA; dolutegravir; weight gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group 1 (Experimental): Delstrigo
  Interventions: Drug: Delstrigo
- Treatment Group 2 (Other): KOCITAF
  Interventions: Drug: KOCITAF

INTERVENTIONS:
Drug: Delstrigo — Treatment Group 1 Participants will receive Doravirine, as part of a fixed-dose oral combination with lamivudine and tenofovir disoproxil fumarate (DOR/3TC/TDF, Delstrigo)tablets which are to be administered orally and once daily.
  Arms: Treatment Group 1
Drug: KOCITAF — Treatment Group 2 Participants will receive dolutegravir, as part of a fixed-dose oral combination with tenofovir alafenamide plus emtricitabine (DTG/TAF/FTC, KOCITAF) tablets which are to be administered orally and once daily.
  Arms: Treatment Group 2

SUMMARY:
This is an open label, randomised, phase 3, two-arm study conducted over 96 weeks.

The study includes a screening period day - 60 to -1, enrolment visit day 0, and a 96-week treatment follow-up period.

Approximately 600 male and female participants infected with HIV-1 eligible for first-line therapy, will be randomly assigned in a 1:1 ratio approximately 300 participants per treatment group to either Treatment Group 1 DOR/3TC/TDF or Treatment Group 2 DTG/TAF/FTC. All medications will be administered in an open label design.

DETAILED DESCRIPTION:
One of the major concerns, voiced by researchers, clinicians, and participants, is that data is severely limited to inform participants with side effects, or those wanting to avoid these side effects, as to evidence-based alternatives. As a result, there are no evidence-based regimens available for participants who have begun experiencing weight gain as a side effect on treatment or wanting to avoid weight gain on initiation of antiretrovirals which is now an almost routine side effect for women or Black participants.

Switching to efavirenz-based regimens, while plausibly associated with weight mitigation in efavirenz slow-metabolizers, is accompanied by unacceptable metabolic, organ and neuropsychiatric side effects in the slow metabolizers likely to experience weight loss. There is minimal data on weight changes for switches from integrase inhibitors and having evidence-based options would dramatically add to treatment possibilities for participants. There is some evidence that the use of TDF and doravirine may mitigate the weight gain seen with TAF/integrase inhibitors combinations.

Doravirine is a compelling replacement for the integrase inhibitors similarly well tolerated, and with a high resistance barrier and better lipid profile as compared to other drugs in the non-nucleoside reverse-transcriptase inhibitor class14. In a recent network meta-analysis, DOR/3TC/TDF was found to exhibit superiority in virological suppression to traditional first line non-DTG containing regimes with more tolerable side effects, and a decrease in severe adverse events.

The DOR/3TC/TDF combination would be a major step forward for current treatment guidelines if found to be equivalent in terms of virological suppression and showed a meaningful difference in weight gain, as well as in cardiometabolic outcomes. This potentially offers clinicians and high risk participants an evidence-based alternative to TAF/integrase inhibitor combinations.

We propose a head-to-head, non-inferiority, randomized study with DTG/TAF/FTC, against a formulation of DOR/3TC/TDF, in antiretroviral-naïve overweight participants, with differences in viral suppression as the primary end points weight gain and metabolic changes-being secondary endpoints of interest at 48 Weeks.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all the following criteria to be enrolled in this study.

* ≥18 years old, male or female.
* Documented laboratory diagnosis of infection with HIV-1 (positive enzyme-linked immunosorbent assay HIV-1 antibody test) at screening, with no baseline DOR resistance (please see Table 2 below).
* Is ART naïve.
* BMI≥ 25 kg/cm2.
* VL >500 copies/ml.
* Must sign an ICF indicating that he or she understands the purpose of, and procedures required for the study and is willing to participate in the study.
* Female participants of childbearing potential (WOCBP) are eligible to participate if willing to use highly effective contraception methods from enrolment, for the duration of the study.

Exclusion criteria:

Participants meeting any of the following criteria will be excluded from the study:

* Is currently participating in any other interventional study or participated in a study with an investigational drug within 60 days of screening.
* Is pregnant, breastfeeding or intends to become pregnant or breastfeed during the study.
* Has active TB co-infection and requires anti-TB treatment.
* Has unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypalbuminaemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones); Child-Pugh C.
* Has pre-existing physical or mental condition (including substance abuse disorder and suicide risk) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Clinically unstable in the investigator's opinion (any pre-existing medical or laboratory abnormalities must be deemed to be stable by the investigator prior to study enrolment).
* Has estimated creatinine clearance <60mL/min per Cockcroft-Gault formula.
* Is taking, and is unable to discontinue, any of the following prohibited medications: carbamazepine, oxcarbazepine, phenobarbital, phenytoin; the antimycobacterial rifampicin, rifapentine; St. John's Wort (Hypericum perforatum); mitotane; enzalutamide; lumacaftor.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The antiretroviral activity of DOR/3TC/TDF compared to DTG/TAF/FTC in the first line treatment, as assessed by the percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 | 48 Weeks
  HIV1-RNA

SECONDARY OUTCOMES:
The antiretroviral activity of DOR/3TC/TDF compared to DTG/TAF/FTC, as assessed by the percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 | 96 Weeks
  HIV-1 RNA
The antiretroviral activity of DOR/3TC/TDF compared with DTG/TAF/FTC, as assessed by the percentage of participants with HIV-1 RNA <200 copies/mL at Week 48 and Week 96 | 48 and 96 Weeks
  HIV-1 RNA
Time to virologic failure (defined as confirmed HIV-1 RNA levels ≥ 1000 copies/mL at week 24 or ≥ 200 copies/mL after week 24) | 24 Weeks
  HIV-1 RNA
The immunologic effect of DOR/3TC/TDF compared with DTG/TAF/FTC, as assessed by the mean change from baseline in CD4+ T-cell count at Week 48 and Week 96 | 48 and 96 Weeks
  CD4-T-cell count
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 96 Weeks
  Adverse events
The effect of DOR/3TC/TDF compared with DTG/TAF/FTC on weight, as assessed by the mean change from baseline to Week 48 and Week 96 | 48 and 96 Weeks
  Weight
The effect on body composition of DOR/3TC/TDF compared with DTG/TAF/FTC, as assessed by the mean change from baseline to Week 48 and Week 96. | 48 and 96 Weeks
  Dual-energy X-ray absorptiometry (DXA) scan
The effect on hematology of DOR/3TC/TDF compared with DTG/TAF/FTC, as assessed by the mean change from baseline to Week 48 and Week 96. | 48 and 96 Weeks
  Full blood count
The effect on lipid profile of DOR/3TC/TDF compared with DTG/TAF/FTC, as assessed by the mean change from baseline to Week 48 and Week 96 | 48 and 96 Weeks
  fasting lipogram
To evaluate the pharmacokinetics of DOR in pregnant women | 96 Weeks
  Peak Plasma Concentration (Cmax)
To evaluate the pharmacokinetics of DOR in pregnant women | 96 Weeks
  Area under the plasma concentration versus time curve (AUC)

OTHER OUTCOMES:
To evaluate the pharmacokinetics of DOR in pregnant women | 96 Weeks
  The observed concentration at 24 hours after dose administration
Number of pregnant women with treatment related adverse events as assessed by (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events v2.1 | 96 Weeks
  Grade 4 AEs which are potentially life-threatening events.
To describe Patient-Reported Outcomes (PROs) for participants who received DOR/3TC/TDF compared with DTG/TAF/FTC overtime | 96 Weeks
  Change in quality of life (QoL) using, defined as the difference in the summary scores obtained from each individual question (higher scores better outcome)
To describe Patient-Reported Outcomes (PROs) for participants who received DOR/3TC/TDF compared with DTG/TAF/FTC overtime | 96 Weeks
  Sleep measurement using the sleep assessment questionnaire the participant answers on a scale of 1 - 10, a score >4 indicates a higher likelihood of insomnia
To describe Patient-Reported Outcomes (PROs) for participants who received DOR/3TC/TDF compared with DTG/TAF/FTC overtime | 96 Weeks
  Food Intake Diary there is no min or max values assessments will be done based upon participant diet
To describe Patient-Reported Outcomes (PROs) for participants who received DOR/3TC/TDF compared with DTG/TAF/FTC overtime | 96 Weeks
  Mental health questionnaire with higher scores means more risk of mental distress, grand total more than 7 requires referrals for mental health assessment by investigator.

CONTACTS AND LOCATIONS:
Overall Officials: JOANA FRANCISCA WOODS, MBBCh, Principal Investigator — Ezintsha Resesarch Centre; SIMISO MANDISA Sokhela, MBBCh, Study Director — Ezintsha Research Centre
Locations (1):
- Ezintsha Research Centre, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately following publication